CLINICAL TRIAL: NCT04306276
Title: Pretreatment With Dienogest in Women With Endometriosis Undergoing in Vitro-fertilization After a Previous Failed Cycle
Status: Completed | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Fabio Barra, Principal Investigator, Ospedale Policlinico San Martino
Other Study IDs: DIENIVF-ENDO
Record Dates: First submitted 2020-03-08; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Endometriosis; Endometriosis Ovary; IVF
Keywords: endometriosis; IVF
MeSH Terms: conditions — Endometriosis | interventions — dienogest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing direct IVF: Patients directly undergo IVF without receiving previous hormonal treatment
- Patients pretreated with DNG: Patients having received a three-month treatment with DNG before undergoing IVF
  Interventions: Drug: Dienogest 2 MG

INTERVENTIONS:
Drug: Dienogest 2 MG — Three-month treatment with DNG (2 mg daily; Visanne, Bayer Pharma, Germany) before IVF
  Groups: Patients pretreated with DNG

SUMMARY:
It is generally assumed that the major causes of in vitro fertilization (IVF) failure in women with endometriosis are diminished ovarian reserve, impaired endometrial receptivity and low quality of embryos. The use of prolonged courses of hormone therapy may play an important role in the strategy of overcoming endometriosis-related infertility. The aim of this study was to evaluate the use of dienogest (DNG) before an IVF cycle in women with endometriosis undergone a previous IVF failed cycle

DETAILED DESCRIPTION:
The primary outcomes of the study are clinical pregnancy rate and live birth rate after reaching 24 week's gestation.

Secondary outcomes of the study are: changes in the diameter and volume of the largest endometrioma, total gonadotropin dose administered, number of mature oocytes collected, number of two-pronuclear (2PN) embryos, number of blastocysts.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of endometriosis at magnetic resonance imaging or transvaginal ultrasonography;
* one failed previous IVF cycle (including failure of frozen embryo transfer);
* basal FSH < 14.0 IU/L;
* antimullerian hormone (AMH) blood level >= 0.5 g/mL;
* normal thyroid-stimulating hormone and prolactin.

Exclusion Criteria:

* history of surgery for endometriosis;
* history of uterine or adnexal surgery;
* use of hormonal therapies for the treatment of endometriosis related pain within 6 months before IVF;
* adenomyosis (magnetic resonance imaging or transvaginal ultrasonography);
* hydrosalpinx;
* submucosal fibroids;
* body mass index (BMI) ≥ 30 kg/m2;
* severe male factor infertility (< 5 million total motile sperm count).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with endometriosis who previously failed one IVF cycle and all resultant frozen embryo transfer
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 8 weeks
Live birth rate after reaching 24 week's gestation | 24 weeks

SECONDARY OUTCOMES:
Total gonadotropin dose administered | During the procedure
Number of mature oocytes collected | During the procedure
Number of two-pronuclear (2PN) embryos | During the procedure
Number of blastocysts. | During the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Barra, MD, PhD, Principal Investigator — IRCCS Ospedale Policlinico San Martino
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided